CLINICAL TRIAL: NCT06821347
Title: NanO2 in Large VessEL Occlusion Stroke (NOVEL): a Multicentre Single-blind, Randomised, Placebo-controlled Blinded Biomarker End-point Clinical Trial of Perfluorocarbon in Acute Ischaemic Stroke Due to Large Vessel Occlusion
Brief Title: NanO2 in Large VessEL Occlusion Stroke (NOVEL)
Acronym: NOVEL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other); NuvOx LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GN21ST331; NIHR151755 (Other Grant/Funding Number: National Institute for Health Research)
Record Dates: First submitted 2025-02-10; First posted 2025-02-12 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-02

CONDITIONS: Stroke Acute
Keywords: acute ischaemic stroke; large vessel occlusion; thrombolysis
MeSH Terms: conditions — Stroke | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Statisticians
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- NanO2 (Experimental)
  Interventions: Drug: NanO2TM
- Placebo (Placebo Comparator)
  Interventions: Other: Sodium Chloride 0.9% Intravenous

INTERVENTIONS:
Drug: NanO2TM — Intravenous NanO2 0.17ml/kg (three doses given over 4.5 hours)
  Arms: NanO2
Other: Sodium Chloride 0.9% Intravenous — Placebo
  Arms: Placebo

SUMMARY:
This is a National Institute for Health Research (NIHR) Efficacy and Mechanism Evaluation (EME) clinical trial aiming to investigate a possible new treatment to limit damage to the brain caused by a stroke. Strokes that are caused by a clot blocking an artery in the brain ('ischaemic' strokes) starve brain tissue of oxygen and nutrients. Over a short period of time without oxygen, this tissue becomes permanently damaged. The trial aims to investigate the effects of a drug that carries extra oxygen, called NanO2, on the amount of brain tissue damage. By carrying extra oxygen to brain tissue NanO2 may allow the tissue to survive for longer. It might be especially useful to prevent further damage happening while treatments to try and open the blocked blood vessel are given. Treatments may include 'clot-busting' drugs, or procedures to physically open a blocked artery. These treatments are very effective, but take time to successfully open the blockage. The study will involve treating people as early as possible after the stroke, and comparing brain scans before and after treatment. Patients diagnosed with a stroke that has occurred within the past 9 hours will be eligible to participate. The study will involve 8-15 hospitals across the UK. Participation in the study will last approximately 90 days. The majority of the study assessments will be during the first 5 days during inpatient hospital stay. There will be a telephone follow-up at 30 days and 90 days post-discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female aged ≥ 18 years
2. Acute ischemic stroke fulfilling perfusion imaging criteria (ischemic core volume < 70 mL, mismatch ratio > 1.8 and mismatch volume > 15 mL using RAPID or equivalent CE-marked software)
3. Eligible for thrombolysis or thrombectomy
4. Intracranial LVO on CTA (occlusion of the terminal ICA, MCA-M1, ≥1 proximal MCA-M2, or proximal posterior cerebral artery (PCA-P1))
5. ≤ 9 hours after last known well (if waking with symptoms, last known well time is calculated as the mid-point between going to sleep and waking)
6. Pre-stroke functional independence (estimated pre-stroke mRS ≤2)
7. NIHSS score ≥ 6 (or NIHSS ≥ 2 if PCA-P1 occlusion) at randomisation

Exclusion Criteria:

1. History of significantly impaired renal eGFR (<30ml/min) or hepatic function (transaminases >3 times upper limit of normal or history of cirrhosis), unstable angina or heart failure (NYHA 3 or 4).
2. Pre-existing lung disease requiring supplemental chronic or intermittent oxygen therapy (NB oxygen therapy given post-stroke is not an exclusion)
3. Previous hypersensitivity reaction to NanO2 excipients and/or compounds similar to NanO2
4. Pregnancy (for women of child-bearing potential a negative pregnancy test will be required prior to randomisation) or breast feeding women.

   Women of child-bearing potential is defined as experienced menarche; AND not undergone successful surgical sterilisation (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy); AND not post-menopausal i.e. amenorrhea for ≥12 consecutive months (without another medical cause)
5. Participation in another CTIMP within preceding 90 days or 5 half-lives of the investigational product, whichever is longer, or previous participation in NOVEL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Volume of penumbral tissue salvaged based on follow-up imaging (diffusion weighted MRI, or non-contrast CT if MRI cannot be obtained) compared with pre-treatment penumbral tissue volume from CT Perfusion. | Baseline to 24hrs

SECONDARY OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS) change from baseline to day 5 | Baseline to Day 5
  The National Institutes of Health Stroke Scale (NIHSS) is a 15-item neurologic examination in stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. Ratings for each item are scored with 3-5 grades with 0 normal, and there is an allowance for untestable items.
NIHSS score change from baseline to 24h | Baseline to 24hrs
  The National Institutes of Health Stroke Scale (NIHSS) is a 15-item neurologic examination in stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. Ratings for each item are scored with 3-5 grades with 0 normal, and there is an allowance for untestable items.
24 hour NIHSS score | Baseline to 24hrs
  The National Institutes of Health Stroke Scale (NIHSS) is a 15-item neurologic examination in stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. Ratings for each item are scored with 3-5 grades with 0 normal, and there is an allowance for untestable items.
Proportion achieving substantial early neurological improvement (NIHSS score reduced by ≥8 points or a score equal to 0 or 1) at 24 hours | Baseline to 24hrs
  The National Institutes of Health Stroke Scale (NIHSS) is a 15-item neurologic examination in stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. Ratings for each item are scored with 3-5 grades with 0 normal, and there is an allowance for untestable items.
Distribution of modified Rankin Scale (mRS) scores at 30 and 90 days | Baseline to Day 30 and Day 90
  The mRS is a hierarchial ordinal scale used to assess disability in stroke trials, with seven discrete levels that range from No Symptoms (mRS=0) to Death (mRS=6)
Proportion achieving independence (mRS score ≤2) at 90 days | Baseline to Day 90
  The mRS is a hierarchial ordinal scale used to assess disability in stroke trials, with seven discrete levels that range from No Symptoms (mRS=0) to Death (mRS=6)
Proportion achieving excellent neurological outcome (mRS score 0-1) at 90 days | Baseline to Day 90
  The mRS is a hierarchial ordinal scale used to assess disability in stroke trials, with seven discrete levels that range from No Symptoms (mRS=0) to Death (mRS=6)
Health-related Quality of Life using the EQ-5D score at 90 days | Baseline to Day 90
  EQ5D is a standardised instrument for use as a measure of health outcome. EQ5D is a descriptive system of health-related quality of life states consisting of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each of which can take one of three responses reflecting severity (no problems / some or moderate problems / extreme problems). Participants are asked to rate their health today using a scale of 0 (worst health imaginable) to 100 (best health imaginable).
Mortality | Baseline to Day 90
Cumulative incidence of Serious Adverse Events at 24h, day 5 and day 90 | Baseline to Day 90

CONTACTS AND LOCATIONS:
Locations (1):
- NHS Greater Glasgow and Clyde, Glasgow, United Kingdom, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing will be facilitated in line with co-sponsor policies. Consent to share non-identifiable data with other researchers will be sought from study participants prior to participation.